CLINICAL TRIAL: NCT05385250
Title: Bone-sparing Chemoradiotherapy for Anal Cancer - A Prospective Phase II Trial Danish Anal Cancer Group Study
Brief Title: Bone-sparing Chemoradiotherapy for Anal Cancer - DACG-II
Acronym: DACG-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karen-Lise Garm Spindler (Other)
Collaborators: Herlev Hospital (Other); Zealand University Hospital (Other); Vejle Hospital (Other)
Responsible Party: Sponsor-Investigator, Karen-Lise Garm Spindler, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DACG-II
Record Dates: First submitted 2022-02-24; First posted 2022-05-23 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Anal Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Anus Neoplasms; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: A phase II prospective observational clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone sparring radiotherapy (Other): Observational arm of bone-sparing radiotherapy
  Interventions: Other: Bone sparring radiotherapy

INTERVENTIONS:
Other: Bone sparring radiotherapy — Observation of late side effects from the pelvic bones after bone-sparring radiotherapy for anal cancer

SUMMARY:
This study proposal includes a prospective clinical trial of bone sparing treatment planning in anal cancer patients. the trial aim to lower the risk of bone damage, while adhering with the constrains to the bowel, bladder and other conventional Organs At Risk, and finally to describe the fraction of pelvic insufficiency fractures in patients treated with optimized radiotherapy.

DETAILED DESCRIPTION:
Patients will receive standard (chemo)-radiotherapy according to national Danish Anal Cancer Group (DACG) guidelines, but the bone-sparing focus will be added to the algorithm for dose-constrains and planning objectives. A bone specific magnetic resonance scan will be performed at 1 year post treatment. Additional substudies include collection of blood samples for translational research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy verified localized squamous cell anal cancer
* Indication for standard (chemo)-radiotherapy with curative intend for anal cancer as per multidisciplinary team decision
* Clinical eligible for standard (chemo)-radiotherapy as per physicians' decision
* Written and oral consent
* Age at least 18 years

Exclusion Criteria:

* Previous pelvic radiotherapy
* Previous systemic therapy with severe bone marrow suppression or hematological diseases
* Hip-replacements
* Contraindications to MRI-scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of PIFs | 1 year
  Rate of pelvic insufficience fractures (PIF) on MRI

SECONDARY OUTCOMES:
Rate of symptomatic PIFs | after 1 and 3 year
  Rate of symptomatic Pelvic insufficiency fractures (PIF)
Rate of toxicity from standard organs at risk (OAR) | after 1 and 3 years
  Rate of physician rated toxicity from standard OAR; bowel, bladder, skin
Predictive and prognostic biomarkers | Pre-treatment, By end of therapy (on average 30 days) and after 1 and 3 years
  Prognostic value of levels of circulating DNA (copies per ML) in blood samples
Patient reported outcomes measures (LARS) | Pretreatment and at 1 and 3 years
  Patient reported outcome measure by LARS (low anterior resection syndrome) scores 1-5
Patient reported outcome measures (FACT-BP) | Pretreatment and after 1 and 3 years
  Patient reported outcome measures by Functional Assessment of Cancer Therapy - Bone Pain score
Quality of Life measures (EORTC) | Pretreatment and after 1 and 3 years
  Quality of Life measures (EORTC)

CONTACTS AND LOCATIONS:
Overall Officials: Karen-Lise G Spindler, DMSc, PhD, Study Chair — Experimental Clinical Oncology, AUH, And Danish Anal Cancer Group, DACG
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No